CLINICAL TRIAL: NCT01361126
Title: A Phase I/II Open-label, Multicenter, Safety and Efficacy Study of a Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) in Subjects With Hemophilia B
Brief Title: A Safety and Efficacy Study of a Recombinant Factor IX in Patients With Severe Hemophilia B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL654_2004; 2010-023793-39 (EudraCT Number)
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — albutrepenonacog alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On-demand (Experimental): The routine prophylactic therapy interval is targeted at every 7 days.
  Interventions: Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein
- Prophylactic (Experimental): On-demand subjects will receive rIX-FP only for the treatment of a bleeding episode.
  Interventions: Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein

INTERVENTIONS:
Biological: Recombinant Coagulation Factor IX Albumin Fusion Protein — Study subjects will receive a single dose of 25IU/kg of rIX_FP for pharmacokinetic analysis. Subjects will then be treated for approximately 5 months. The treatment dose will be based on the subject's PK profile and the subject's bleeding phenotype.
  Other Names: CSL654

SUMMARY:
This study will examine the safety and efficacy of a Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) for the control and prevention of bleeding episodes in subjects who have previously received factor replacement therapy for hemophilia B. The study consists of a screening period, a pharmacokinetic (PK) period, followed by approximately a 5 month treatment period. Subjects will receive weekly routine prophylactic therapy and on-demand treatment for bleeding episodes. In addition, subjects who are not on routine factor replacement therapy prior to the study will receive only on-demand treatment for bleeding episodes.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, 12 to 65 years old
* Severe hemophilia B (FIX activity of ≤ 2%)
* Subjects who have received FIX products (plasma-derived and/or recombinant FIX) for > 150 exposure days (EDs)
* No history of FIX inhibitor formation, no detectable inhibitors at Screening and no family history of inhibitors against FIX
* Written informed consent for study participation obtained before undergoing any study specific procedures

Exclusion Criteria:

* Known hypersensitivity to any FIX product or hamster protein
* Known congenital or acquired coagulation disorder other than congenital FIX deficiency
* HIV positive subjects with a CD4 count < 200/mm3
* Low platelet count, abnormal kidney function, or liver disease
* On-demand subjects experiencing less than 12 or 6 non-trauma induced bleeding episodes requiring treatment with a FIX product during the previous 6 or 3 months, respectively
* Planned major surgical intervention during the study period

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Jacobs, MD, Study Director — CSL Behring
Locations (2):
- Study Site, Sofia, Bulgaria
- Study Site, Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 17 subjects were screened and enrolled in the study. Fifteen subjects participated in the pharmacokinetic (PK) evaluation period and were administered a dose of 25 IU/kg rIX-FP. Two subjects did not participate in the PK evaluation period because PK data for these 2 subjects were available from the previous phase 1 study (CSL654_2001).
Groups:
- Prophylactic: For the PK evaluation, subjects received a single intravenous (IV) infusion of Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) at a dose of 25 IU/kg. After completion of the PK evaluation period, subjects entered the treatment period and were administered a single IV infusion of rIX-FP once a week at a dose of 15 to 35 IU/kg, or at a dose determined by the investigator. The dose was adjusted up to 75 IU/kg to maintain the trough FIX activity level > 1% between infusions.
- On-demand: For the PK evaluation, subjects received a single IV infusion of rIX-FP at a dose of 25 IU/kg. After completion of the PK evaluation period, subjects entered the treatment period and were administered 1 or more IV infusions of rIX-FP at a dose of at least 25 IU/kg to treat minor, moderate or major bleeding episodes. The dose of rIX-FP was calculated by the investigator.
Period: Overall Study
Arm/Group | Prophylactic | On-demand
Started | 13 | 4
Completed | 13 | 2
Not Completed | 0 | 2
Not completed — Sponsor decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Prophylactic: For the PK evaluation, subjects received a single IV infusion of rIX-FP at a dose of 25 IU/kg. After completion of the PK evaluation period, subjects entered the treatment period and were administered a single IV infusion of rIX-FP once a week at a dose of 15 to 35 IU/kg, or at a dose determined by the investigator. The dose was adjusted up to 75 IU/kg to maintain the trough FIX activity level > 1% between infusions.
- Total: Total of all reporting groups
Arm/Group | Prophylactic | On-demand | Total
Number analyzed (Participants) | 13 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (9.4) | 35.8 (9.7) | 26.1 (10.7)
Age, Customized [Number; unit: participants]
  < 18 years | 3 | 0 | 3
  ≥ 18 years | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-related Adverse Events
Description: The causal relationship of each adverse event to rIX-FP was assessed by the Investigator.
Time Frame: Approximately 20 weeks
Population: Safety Population
Measure: Number; unit: participants
Groups:
- All Subjects: Subjects received rIX-FP as prophylactic treatment once a week or on-demand to treat bleeding episodes administered by IV infusion for 20 weeks.
Arm/Group | All Subjects
Number analyzed (Participants) | 17
participants | 0

2. Primary Outcome: Number of Subjects With Inhibitors Against Factor IX (FIX)
Description: The presence of inhibitors against FIX was assessed by the central laboratory by a FIX potency assay. To quantify anti-FIX neutralizing antibodies, the Bethesda assay with the Nijmegen modification was used, and the results expressed as Bethesda Units per mL (BU/mL). A positive inhibitor test is >=0.6 BU/mL.
Time Frame: Baseline, Day 10 and Weeks 4, 12 and 20
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 17
participants | 0

3. Primary Outcome: Number of Subjects Who Developed Antibodies to rIX-FP
Description: Antibodies against rIX-FP were detected using a direct binding enzyme-linked immunosorbent assay (ELISA).
Time Frame: Pre-dose, Day 10 and Weeks 4, 12, and 20
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 17
participants | 0

4. Secondary Outcome: Area Under the Curve to the Last Sample With Quantifiable Drug Concentration (AUC0-t) After a Single Dose of rIX-FP
Description: The plasma concentrations of rIX-FP were measured as FIX activity using a validated, 1-stage assay in a central laboratory for a quantification range from 0.25 to 150% (or 0.25 IU/dL to 150 IU/dL). The PK population comprised all subjects who received at least 1 dose of rIX-FP and for whom a sufficient number of analyzable PK samples had been obtained in order to permit the evaluation of the PK profile of rIX-FP, and who did not receive a dose of rIX-FP or any other FIX product for the treatment of a bleed during the PK sampling period.
Time Frame: Pre-dose and up to 14 days after rIX-FP infusion.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*IU/dL
Groups:
- Prophylactic; On-demand: For the PK evaluation, subjects received a single IV infusion of rIX-FP at a dose of 25 IU/kg.
Arm/Group | Prophylactic | On-demand
Number analyzed (Participants) | 10 | 3
h*IU/dL | 2915 (11.3) | 2960 (12.4)

5. Secondary Outcome: Half-life (t1/2) of a Single Dose of rIX-FP
Time Frame: Pre-dose and up to 14 days after infusion
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Prophylactic | On-demand
Number analyzed (Participants) | 10 | 3
hours | 77.7 (25.2) | 138 (37.1)

6. Secondary Outcome: Incremental Recovery of rIX-FP at 30 Minutes Following Infusion of rIX-FP
Description: Incremental recovery (IU/mL/IU/kg) is defined as FIX activity (IU/mL) obtained 30 minutes following infusion, per dose of (IU/kg) infusion. FIX activity was measured at a central laboratory using validated one-stage clotting method.
Time Frame: 30 minutes after infusion
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/dL/IU/kg
Arm/Group | Prophylactic | On-demand
Number analyzed (Participants) | 10 | 3
IU/dL/IU/kg | 1.47 (8.2) | 1.35 (4.9)

7. Secondary Outcome: Clearance of a Single Dose of rIX-FP
Time Frame: Pre-dose and up to 14 days after rIX-FP infusion
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Prophylactic | On-demand
Number analyzed (Participants) | 10 | 3
mL/h/kg | 0.749 (14.0) | 0.699 (10.6)

8. Secondary Outcome: Breakthrough Bleeding Events
Description: Number of breakthrough bleeding events (spontaneous bleeding events) requiring treatment per subject in subjects receiving prophylactic treatment regimen with rIX-FP
Time Frame: Week 9 to approximately Week 20
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Events per subject
Arm/Group | Prophylactic
Number analyzed (Participants) | 13
Events per subject | 0.2 (0.38)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- All Subjects: Subjects received rIX-FP administered by IV infusion as prophylactic treatment once a week or on demand to treat bleeding episodes for 20 weeks.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 14/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (11)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (4)
Pharyngitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Injection site swelling (General disorders) | 1 (3)
Injection site erythema (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.